CLINICAL TRIAL: NCT00576745
Title: Comparison Of The 3M Surgical Skin Closure System To The Standard Vicryl Suture Closure Of Sternotomy Incisions
Brief Title: A Comparison Of The 3M TM S Surgical Skin Closure System To The Standard Vicryl Suture Closure of Sternotomy Incisions During Cardiac Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: American Heart Association (Other)
Responsible Party: Principal Investigator, Harold L. Lazar MD, Professor of Cardiothoracic Surgery, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-26298
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Wound Infection
Keywords: Sutures
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Vicryl Suture (Active Comparator): Patients will have their incision closed with vicryl suture
  Interventions: Procedure: Vicryl Suture
- 2 Steri-Strips (Experimental): Patients will have their incisions closed with 3M Surgical-Strips
  Interventions: Device: 3M TM S Surgical Skin Closure System

INTERVENTIONS:
Procedure: Vicryl Suture — A 4-0 vicryl suture will be used to close the subcuticular layer
  Arms: 1 Vicryl Suture
Device: 3M TM S Surgical Skin Closure System — These steri-strips will be applied to close the skin in this cohort of patients
  Arms: 2 Steri-Strips

SUMMARY:
Following closure of surgical incisions, wounds may develop redness, swelling, and drainage which may result in increased pain and infection. This study will test to hypothesis that using the 3M TM S Surgical Skin Closure System will reduce the incidence of pain, redness, swelling, and infections in a group of patients undergoing a mediastinotomy incision used for open heart surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing mediastinotomy for cardiac surgical procedures

Exclusion Criteria:

Patients with:

* Allergies to skin adhesives
* Known keloid formation
* Prior sternotomies
* Conditions making them not candidates for vicryl skin closure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-09; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Incidence of erythema | 30 days following surgery

SECONDARY OUTCOMES:
Incidence of infection | 30 days following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Harold L Lazar MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Result] Lazar HL, McCann J, Fitzgerald CA, Cabral HJ. Adhesive strips versus subcuticular suture for mediansternotomy wound closure. J Card Surg. 2011 Jul;26(4):344-7. doi: 10.1111/j.1540-8191.2011.01257.x. Epub 2011 May 9. PMID 21554389